CLINICAL TRIAL: NCT00233857
Title: Auricular Acupuncture Versus Placebo (Sham Acupuncture) for Postoperative Pain Relief After Ambulatory Knee Arthroscopy - a Randomized Controlled Trial
Brief Title: Auricular Acupuncture for Pain Relief After Ambulatory Knee Arthroscopy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: III UV 23/03
Record Dates: First submitted 2005-10-05; First posted 2005-10-06 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2011-02

CONDITIONS: Postoperative Pain
Keywords: Acute pain; postoperative pain; auricular acupuncture
MeSH Terms: conditions — Pain, Postoperative; Acute Pain | interventions — Acupuncture, Ear

INTERVENTIONS:
Procedure: Auricular acupuncture

SUMMARY:
The aim was to investigate whether auricular acupuncture is superior to sham acupuncture in relief of acute postoperative pain and in reduction of analgesics consumption on demand and their side effects in patients after ambulatory knee arthroscopy

ELIGIBILITY:
Inclusion Criteria:

1. Patients with an American Society of Anesthesiologists physical status of I to II scheduled for ambulatory knee arthroscopy under general anesthesia.
2. Surgery time does not exceed 60 minutes.
3. Patients without previous opioid and/or psychiatric medication.
4. Patients ranged 16-65 years old.
5. Patients able to use Visual Analogue Scale-100 for pain intensity measurement.
6. Patients who have given informed consent.

Exclusion Criteria:

1. Pregnant or nursing females.
2. Recidivist alcoholics and/or patients with history of psychiatric disease.
3. Local or systemic infection.
4. Age < 16 and > 65 years.
5. Surgery time more than 60 minutes.
6. Inability to use Visual Analogue Scale-100.
7. Patients consumed opioid medication before surgery.
8. Patients with prosthetic or damaged cardiac valves (s. Potential risks)
9. Patients who are unable to understand the consent form.

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120
Dates: Start 2003-08; Primary Completion 2004-07 (Actual); Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Postoperative ibuprofen requirement after the surgery

SECONDARY OUTCOMES:
Pain intensity assessed by patients on VAS-100 ; total piritramide requirement in anesthesia recovery room; incidence of analgesia-related side effects

CONTACTS AND LOCATIONS:
Overall Officials: Taras I. Usichenko, Assistant Professor, Principal Investigator — Anesthesiology and Intensive Care Medicine Department, Ernst Moritz Arndt University of Greifswald, Germany
Locations (1):
- Anesthesiology and Intensive Care Medicine Department, University of Greifswald, Germany, Greifswald, Germany